CLINICAL TRIAL: NCT01469221
Title: A Phase 3 International, Double-Bind Trial Evaluating Efficacy and Safety of Multiple Instillations of Intravesical Apaziquone vs. Placebo in Patients With Low-Intermediate Risk Non-Muscle Invasive Bladder Cancer (NMIBC)
Brief Title: Efficacy and Safety Study of Apaziquone vs. Placebo in Patients With Non-Muscle Invasive Bladder Cancer (NMIBC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business reason
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-1012; 2011-003517-42 (EudraCT Number)
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-10

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Non-Muscle Invasive Bladder Cancer; NMIBC; Apaziquone; EOquin; GU Cancer; TURBT
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — apaziquone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apaziquone (Experimental): Apaziquone (4 mg in 40 mL)
  Interventions: Drug: Apaziquone
- Placebo (Placebo Comparator): Matching placebo (40 mL)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apaziquone — 6 weekly multi-instillation of Apaziquone 4 mg in 40 mL
  Other Names: EoQuin; EO9
  Arms: Apaziquone
Drug: Placebo — 6 weekly multi-instillation of matching placebo in 40mL
  Arms: Placebo

SUMMARY:
This is an international, multicenter, double-blind, placebo-controlled, randomized study. All eligible patients entering the open label phase of the study will receive a single immediate instillation of apaziquone (4 mg in 40 mL diluent), post transurethral resection-bladder tumor (TURBT). Following Central Pathology review of histology and Double Blind Phase qualification, patients with confirmed eligibility will be randomized to receive either 6 weekly intravesical instillations of apaziquone or matching placebo and undergo cystoscopic and safety assessments every 3 months for 24 months. Patients with histologic evidence of recurrent disease during the study will be treated according to current treatment guidelines or local standard of care. Safety and efficacy assessments will be performed at 3 month intervals for all randomized patients throughout the study. Patients who receive single dose of apaziquone immediately following TURBT and are not eligible for randomization will be followed for 3 months by cystoscopic exam and safety assessments.

ELIGIBILITY:
Inclusion Criteria (for Open Label):

1. Has the patient given written informed consent and is the patient willing and able to abide by the protocol?
2. Is the patient 18 years old or above?
3. If the patient is a female of childbearing potential, is she using an acceptable/effective method of contraception?
4. Does the female patient of childbearing potential have a negative serum pregnancy test at screening?
5. Does the patient with clinically apparent primary or recurrent low grade Ta NMIBC have :

   * multiple tumors (2-7)
   * No single Tumor > 3 cm
   * No history / evidence of Tis

   Or does the patient with clinically apparent primary or recurrent high grade Ta NMIBC have:
   * A single tumor that is ≤ 3 cm
   * No history / evidence of Tis
6. Is the patient able to retain bladder instillations for a minimum of 60 minutes (± 6 minutes)?
7. Did the patient have upper urinary tract evaluation to exclude urothelial carcinoma, hydronephrosis or renal cell carcinoma or other renal cancers in the 6 months prior to study screening?
8. Is patient's urethra (including prostatic urethra in men) endoscopically free of any visible TCC?
9. For patients with recurrent tumor, did the patient have at least a 6-month cystoscopically-confirmed tumor-free interval between the last tumor recurrence and the time of screening?
10. Has the male patient with a prostate specific antigen (PSA) between 4 and 10 ng/mL had a diagnostic evaluation that reasonably excludes the diagnosis of prostate cancer in the opinion of the Investigator?

Exclusion Criteria (for Open Label):

1. Has the patient received any previous pelvic radiotherapy (includes external beam and/or brachytherapy)?
2. Has the patient ever received apaziquone?
3. Has the patient received an induction course (completed 5 of 6 scheduled weekly instillations) of intravesical BCG (± interferon) with the last dose given less than 12 months ago?
4. Has the patient had any prior intravesical chemotherapy, exclusive of single-dose adjuvant intravesical chemotherapy immediately post-TURBT?
5. Does the patient have a history of urinary retention or a post void residual ≥ 250 cc by bladder scan or ultrasound (post void residual test may be repeated up to 3 times)?
6. Does the patient have or has the patient had any bladder tumor with histology other than transitional cell carcinoma?
7. Does the patient have or has the patient had micro-papillary transitional cell carcinoma?
8. If the patient has recurrent papillary disease of the bladder, has the pathology been anything other than pTa in the past?
9. Does the patient have an active urinary tract infection confirmed by culture or a documented history of recurrent UTI (≥ 6 for females and ≥2 for males per year) in the prior 2 years?
10. Does the patient have a bleeding disorder or a screening platelet count < 50 x 109/L?
11. Does the patient have a screening hemoglobin < 10 g/dL?
12. Does the male patient have a screening serum PSA > 10 ng/mL?
13. Does the patient have a history of Acquired Immunodeficiency Syndrome or HIV positive?
14. Does the patient have a condition or a concurrent severe and/or uncontrolled medical or psychiatric disease (e.g., uncontrolled diabetes, decompensated congestive heart failure, myocardial infarction within 6 months of study, unstable and uncontrolled hypertension, or an active uncontrolled infection), which could compromise participation, compliance with scheduled visits and/or completion of the study?
15. Has the patient participated in an investigational protocol within the past 90 days?
16. Is the patient pregnant or breast feeding?
17. Does the patient have a life expectancy of <3 years?
18. Has the patient had any other malignancy or received therapy for any malignancy in the last five years except

    * non-melanoma skin tumors
    * stage 0 (in situ) cervical carcinoma
    * undetectable PSA for ≥1 year following definitive therapy for localized prostate cancer?
19. Does the patient have documented vesicoureteral reflux or an indwelling ureteral stent?
20. Does the patient have tumor in a bladder diverticulum?
21. Does the patient have a known allergy to red color food dye?

Double-Blind Phase Inclusion Criteria

1. Was all visible tumor resected at the initial TURBT?
2. Does Central Pathology review of the patient's bladder tumor confirm:

   * Low grade Ta disease for multiple tumors (2 - 7) or
   * High Grade Ta disease for single tumor
   * No microscopic evidence of lymphovascular invasion and/or evidence of tumor thromboemboli

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Show-Li Sun, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (29):
- United States (7):
  - Tower Research Institute, Los Angeles, California
  - Department of Urology, University of Miami Miller School of Medicine, Miami, Florida
  - Somerset Urological Associates, PA, Somerville, New Jersey
  - Associated Medical Professionals of New York, PLLC, Oneida, New York
  - Male and Female Urology, Staten Island, New York
  - Associated Medical Professionals of New York, PLLC, Syracuse, New York
  - Alliance Urology Specialists, Greensboro, North Carolina
- Czechia (2):
  - Nemocnice Jablonec nad Nisou, Urologické oddělení, Jablonec nad Nisou
  - Fakultní Thomayerova nemocnice s poliklinikou Urologické oddělení, Prague
- Poland (16):
  - Szpital Miejski im. Prof. E. Michałowskiego, Katowice
  - CenterMed Kraków sp z o.o., Krakow
  - Niepubliczny Zakład Opieki Zdrowotnej-Centrum Medyczne Szpital Świętej Rodziny sp z o.o., Lodz
  - Wojewódzki Szpital Specjalistyczny im. Stefana Kardynała Wyszyńskiego Samodzielny Publiczny Zakład Opieki Zdrowotnej w Lublinie, Oddział Urologii i Onkologii Urologicznej, Lublin
  - Nieubliczny Zakład Opieki Zdrowotnej Europejskie Centrum Zdrowia Otwock im. Fryderyka Chopina Nieubliczny Zakład Opieki Zdrowotnej, Otwock
  - Niepubliczny Zakład Opieki Zdrowotnej Pabianickie Centrum Medyczne, Pabianice
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej, Wojewódzki Szpital Specjalistyczny nr 3, Rybnik
  - Wojewódzki Szpital Specjalistyczny W Siedlcach, Siedlce
  - Pomorska Akademia Medyczna, Szczecin
  - Wojewódzki Szpital Specjalistyczny im Janusza Korczaka, Słupsk
  - Centrum Medycznego Kształcenia Podyplomowego, Samodzielny Publiczny Szpital Kliniczny im. Prof. W. Orłowskiego, Warsaw
  - Wojskowy Instytut Medyczny, Centralny Szpital Kliniczny MON, Warsaw
  - Szpital Bielański im. ks. J. Popiełuszki Samodzielny Publiczny Zakład Opieki Zdrowotnej, Warsaw
  - Szpital Kliniczny Dzieciątka Jezus - Centrum Leczenia Obrażeń, Warsaw
  - Międzyleski Szpital Specjalistyczny w Warszawie Oddział Urologii, Warsaw
  - Wojewódzki Szpital Specjalistyczny we Wrocławiu, Ośrodek Badawczo Rozwojowy, Wroclaw
- Slovakia (4):
  - Univerzitná nemocnica L. Pasteura Košice Univerzitná nemocnica L. Pasteura Košice, Košice
  - Univerzitná nemocnica Martin Urologická klinika, Martin
  - Fakultná nemocnica s poliklinikou J. A. Reimana Prešov Urologická klinika, Prešov
  - Fakultná nemocnica s poliklinikou Žilina Urologické oddelenie, Žilina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients 1) meeting Open Label Phase and Double Blind Phase inclusion and exclusion criteria, including confirmed histology based on Central Pathology Review, and 2) has eligibility packet approved by Sponsor, are randomized in a 1:1 fashion to receive 6 weekly instillations of apaziquone or matching placebo.
Groups:
- Placebo: 6 weekly multi-instillation of matching placebo in 40 mL
- Open Label-Apaziquone: Single dose of Apaziquone 4 mg in 40 mL
Period: Open Label Phase
Arm/Group | Apaziquone | Placebo | Open Label-Apaziquone
Started | 0 | 0 | 47
Completed | 0 | 0 | 44
Not Completed | 0 | 0 | 3
Period: Double Blind Phase
Arm/Group | Apaziquone | Placebo | Open Label-Apaziquone
Started | 14 | 17 | 0
Completed | 0 | 0 | 0
Not Completed | 14 | 17 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Sponsor Terminate Study | 12 | 16 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apaziquone | Placebo | Total
Number analyzed (Participants) | 14 | 17 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 14
  >=65 years | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (9.9) | 63.6 (9.2) | 65.7 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 8 | 11 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 14 | 17 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 17 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Recurrence
Description: Time from randomization to the date of first histologically confirmed recurrence of bladder cancer
Time Frame: 24 Months
Population: Patients who were in the Double Blind Phase
Measure: Median (Full Range); unit: months
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 14 | 17
months | NA [1.5 to 1.5] — only 1 patient recurred, median time to recurrence not reached | 8.5 [2.5 to 8.5]

2. Secondary Outcome: 2-Year Recurrence Rate
Description: Proportion of patients with recurrence at or before 24 months
Time Frame: 24 Months
Population: Patients who were in the Double Blind Phase
Measure: Count of Participants; unit: Participants
Arm/Group | Apaziquone | Placebo
Number analyzed (Participants) | 14 | 17
Participants | 1 | 6

ADVERSE EVENTS:
Arm/Group | Apaziquone | Placebo | Open Label-Apaziquone
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/17 | 0/47
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/17 | 2/47
Other Adverse Events (participants affected / at risk) | 6/14 | 11/17 | 23/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apaziquone (N=14) | Placebo (N=17) | Open Label-Apaziquone (N=47)
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apaziquone (N=14) | Placebo (N=17) | Open Label-Apaziquone (N=47)
Cystitis (Infections and infestations) | 0 | 3 | 3
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 2 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 1 | 2
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No